CLINICAL TRIAL: NCT06187740
Title: A Phase I Dose Escalation Study of Thoracic Consolidation Radiotherapy for Extensive-stage Small Cell Lung Cancer Patients Treated With Chemo-immunotherapy
Brief Title: Thoracic Consolidation Radiotherapy for ES-SCLC Treated With Chemo-immunotherapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Chief physician, Department of Radiation Oncology, Fudan University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ES-SCLC-TRT
Record Dates: First submitted 2023-12-17; First posted 2024-01-03 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Small Cell Lung Cancer Extensive Stage
Keywords: small cell lung cancer; chemotherapy; immunotherapy; thoracic radiotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Intervention Model Description: Initial dose of 30 Gy in 10 fractions (3 patients, Arm 1). Dose escalation will start after acceptable safety was observed, 35 Gy/10Fx (3 patients, Arm 2), 40 Gy/10Fx (22 patients, Arm 3).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Starting Dose, Arm 1 (Experimental): For ES-SCLC patients who completed first-line four-cycle chemo-immunotherapy, and was evaluated to have any response to treatment. Thoracic radiotherapy is administered to treat residual thoracic lesions during immunotherapy maintenance phase. Thoracic radiotherapy should begin within 42 days after the end of the last chemotherapy at an initial dose of 30 Gy in 10 fractions (3 patients).
  Interventions: Radiation: thoracic radiotherapy
- Dose escalation 1, Arm 2 (Experimental): Dose escalation will start after acceptable safety was observed, first at: 35 Gy/10 Fx (3 patients). Radiotherapy was administered between two immunotherapy doses (3 weeks interval) to avoid thoracic radiotherapy on the same day with immunotherapy.
  Immunotherapy was maintained until disease progression or the investigator 's judgment there was no further benefit from immunotherapy, patient died, intolerable toxicity developed. Toxicities were assessed periodically during the study. Local radiotherapy is permitted for symptomatic brain/bone metastases.
  Interventions: Radiation: thoracic radiotherapy
- Dose escalation 2, Arm 3 (Experimental): Dose escalation will continue after acceptable safety was observed in the previous dose gourp, at: 40 Gy/10 Fx (22 patients). Radiotherapy was administered between two immunotherapy doses (3 weeks interval) to avoid thoracic radiotherapy on the same day with immunotherapy.
  Immunotherapy was maintained until disease progression or the investigator 's judgment there was no further benefit from immunotherapy, patient died, intolerable toxicity developed. Toxicities were assessed periodically during the study. Local radiotherapy is permitted for symptomatic brain/bone metastases.
  Interventions: Radiation: thoracic radiotherapy

INTERVENTIONS:
Radiation: thoracic radiotherapy — Thoracic radiotherapy should begin within 42 days after the end of the last chemotherapy at an initial dose of 30 Gy in 10 fractions (3 patients).
  Dose escalation will start after acceptable safety was observed, first at: 35 Gy/10 Fx(3 patients), then to the next dose group: 40 Gy/10 Fx(22 patients). Radiotherapy was administered between two immunotherapy doses (3 weeks interval) to avoid thoracic radiotherapy on the same day with immunotherapy.

SUMMARY:
This study intends to recruit ES-SCLC patients with response to standard first-line chemo-immunotherapy to assess the safety of receiving different doses of consolidative thoracic radiotherapy.

DETAILED DESCRIPTION:
Approximately two-thirds of Small-cell lung cancer (SCLC) patients are in the extensive stage (Extensive-Stage SCLC, ES-SCLC) at the time of diagnosis, and the 5-year survival rate of these patients is less than 5%. Before the immunotherapy era, the standard first-line treatment for ES-SCLC had been platinum-based chemotherapy regimens combined with etoposide.

Since treatment failure patterns revealed high probability of residual thoracic disease and high risk of progression of thoracic lesions after ES-SCLC chemotherapy, previous studies suggest that thoracic consolidation radiotherapy in ES-SCLC patients who are sensitive to first-line chemotherapy can reduce the risk of thoracic recurrence and improve overall survival time. Slotman et al. further conducted a phase III randomized controlled clinical study to explore the application of thoracic consolidation radiotherapy in ES-SCLC (CREST study). The CREST study results showed that in ES-SCLC patients who responded to chemotherapy and had residual thoracic lesions, thoracic residual lesion radiotherapy (30 Gy/1 0Fx) combined with prophylactic brain radiotherapy could reduce the risk of thoracic recurrence by 50% and increase the 2-year survival rate from 3% to 13%.

With the advent of the era of immunotherapy, the IMpower133 trial showed that the combination of atezolizumab and chemotherapy prolonged the median overall survival time of ES-SCLC patients compared with the chemotherapy alone group. In the CASPIAN study, the combination of dulvumab and chemotherapy also resulted in a survival benefit. The ASTRUM-005 study using PD-1 monoclonal antibody Serplulimab in combination with chemotherapy also achieved prolonged overall survival.

Although the overall median survival of ES-SCLC is prolonged after immunotherapy in combination with chemotherapy, patients who truly achieve long-term survival are still limited, with a 3-year OS rate of about 15% - 20%. Accordingly, it is necessary to explore effective methods to combine radiotherapy and maximize the benefit population of immunotherapy in ES-SCLC.

Failure pattern analysis revealed that, consistent with the era of non-immunotherapy, the main progression phenotype in patients receiving first-line chemotherapy + immunotherapy remained thoracic progression, suggesting that sequential thoracic consolidation radiotherapy is still likely to achieve clinical benefit in ES-SCLC patients receiving chemo-immunotherapy.

Immunotherapy combined with concurrent chemoradiotherapy has shown good safety and survival benefit in limited-stage SCLC. In non-small cell lung cancer (NSCLC), the safety of sequential immunotherapy after thoracic chemoradiotherapy has also been verified. However, there is a lack of prospective studies to investigate the safety of sequential thoracic consolidation radiotherapy after first-line immunochemotherapy in ES-SCLC patients.

At present, the widely used ES-SCLC thoracic consolidation radiotherapy regimen is based on the 30 Gy/1 0Fx dose fractionation of CREST study. At the same time, it has been shown that increasing the dose of single radiotherapy within a certain range helps to increase the production of immunogenic death by tumor cells, that is, more tumor-specific antigens that can be recognized by the immune system are produced during the induction of tumor cell death. Therefore, this study intends to perform a dose escalation study based on 30 Gy/10Fx dose fractionation and assess the safety of this treatment mode.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

1. age ≥ 18 years;
2. ECOG performance status score 0-2 points;
3. pathologically confirmed small cell lung cancer;
4. complete baseline imaging data (including brain enhanced MRI/CT, PET-CT or chest enhanced CT + bone scan + neck and abdominal B ultrasound/CT) before first-line treatment;
5. stage extensive-stage SCLC at initial diagnosis, and first-line treatment received standard platinum-based doublet chemotherapy combined with immunotherapy (PD-1 or PD-L1) for at least 4 cycles after the efficacy assessment of SD or PR (residual lesions assessed by chest CT);
6. no history of other malignancies;
7. reproductive age male/female agreed to contraception during the trial (surgical ligation or oral contraceptives/intrauterine devices + condom contraception);
8. life expectancy ≥ 3 months
9. 1 week before enrollment, the investigator judged that the patient could continue immune maintenance therapy at the same time, And the organ function level meets the following criteria:

1) bone marrow function: hemoglobin ≥ 80 g/L, white blood cell count ≥ 4.0 * 10 ^ 9/L or neutrophil count ≥ 1.5 * 10 ^ 9/L, platelet count ≥ 100 * 10 ^ 9/L; 2) liver: serum total bilirubin level ≤ 1.5 times the upper limit of normal, when serum total bilirubin level > 1.5 times the upper limit of normal direct bilirubin level must be ≤ the upper limit of normal,Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times of the upper limit of normal; serum albumin ≥ 27 g/L; 3) Kidney: serum creatinine level < 1.5 times of the upper limit of normal or creatinine clearance ≥ 50 ml/min, urea nitrogen ≤ 200 mg/L; 10.Patients must have the ability to understand and voluntarily sign an informed consent form.

Exclusion Criteria:

1. baseline pathological examination found mixed with non-small cell lung cancer components;
2. patients who had used any anti-tumor therapy before the diagnosis of ES-SCLC;
3. patients who had received anti-tumor therapy other than standard chemotherapy + immunotherapy regimen;
4. patients who had PD assessed by chemotherapy combined with immunotherapy efficacy;
5. patients who had no residual thoracic lesions (lung, mediastinal and supraclavicular metastatic lymph nodes, thoracic efficacy CR) on chest enhanced CT during efficacy assessment;
6. patients with severe immune-related toxicities after treatment;
7. symptomatic interstitial lung disease or active infection/non-infectious pneumonia;
8. patients who required long-term use of cortisol or immunosuppressive agents;
9. allergic to PD-1 or PD-L1 monoclonal antibody immunotherapy or other causes of inability to perform immune maintenance therapy;
10. lactating or pregnant women;
11. patients with severe autoimmune diseases: active inflammatory bowel disease (including Crohn 's disease, ulcerative colitis), rheumatoid arthritis, scleroderma, systemic lupus erythematosus, autoimmune vasculitis (such as Wegener' s granulomatosis), etc.;
12. researchers believe that physical examination or clinical trials may interfere with the results or increase the risk of treatment complications, or other uncontrollable diseases;
13. patients with mental illness, substance abuse, social problems affecting compliance are not enrolled after the doctor 's review.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related dose-limiting toxicities (DLTs) | 90 days after the start of thoracic consolidation radiotherapy in enrolled patients
  The proportion of the number of cases with DLTs associated with the study design treatment to the total evaluable number of cases was assessed according to CTCAE 5.0 criteria.
  Definition of dose-limiting toxicities (DLTs): Grade 3 or higher non-hematological/laboratory abnormalities reported events that may or definitely be associated with the combination of immunotherapy and thoracic consolidation radiotherapy as judged by the investigator, or Grade 4 or higher hematological/laboratory abnormalities reported.

SECONDARY OUTCOMES:
Incidence of all dose limiting toxicities (DLTs): | 90 days after the start of thoracic consolidation radiotherapy in enrolled patients
  Incidence of all dose limiting toxicities (DLTs): The proportion of cases with DLTs (whether judged treatment-related or not) as assessed by CTCAE 5.0 criteria compared with the total evaluable cases

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No